CLINICAL TRIAL: NCT02473874
Title: Spectral Comparison Between Spatially Modulated Quantitative Spectroscopy and Polarization-Sensitive Hyperspectral Multimode Dermoscopy for the Purpose of Skin Compositional Analysis
Brief Title: Comparison Imaging System Between Spatially Modulated Quantitative Spectroscopy and Skin Spect Dermoscopy
Status: Withdrawn | Type: Observational
Why Stopped: Not NIH defined clinical trial study.
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Kristen Kelly, M.D., Professor of Dermatology and Surgery, University of California, Irvine
Other Study IDs: 20151791
Record Dates: First submitted 2015-06-05; First posted 2015-06-17 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Melanocytic Nevus
MeSH Terms: conditions — Nevus, Pigmented

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Skin Spect dermoscope: Skin mole
  Interventions: Device: Skin Spect dermoscope
- Spatially modulated quantitative: Skin mole
  Interventions: Device: Spatially modulated quantitative

INTERVENTIONS:
Device: Skin Spect dermoscope — Skin imaging
  Groups: Skin Spect dermoscope
Device: Spatially modulated quantitative — Skin imaging
  Groups: Spatially modulated quantitative

SUMMARY:
The purpose of this study is to obtain skin spectroscopic data from two imaging systems.

Comparison groups:

* Skin Spect dermoscope
* Spatially modulated quantitative spectrometer

DETAILED DESCRIPTION:
The researcher can compare the spectroscopic data from the two systems as well as the relative concentrations of melanin, oxy- and deoxy- hemoglobin calculated from the measurements.

Skin Spect can measure larger area of skin, whereas Spatially modulated quantitative spectrometer is a point-based measurement.Therefore, larger nevi will require multiple Spatially modulated quantitative spectrometer measurements for comparison with corresponding sub-regions of the larger Skin Spect measurements. Only sub-regions of the image data from Skin Spect that match the locations Spatially modulated quantitative spectrometer acquired data will be used in this correlation study.

This researcher ensure that the spectral data collected by the two instruments are collected from the same spatial locations, should lesion heterogeneity be present.

ELIGIBILITY:
Inclusion Criteria:

* Skin lesion a mole located on flat surface of the body

Exclusion Criteria:

* Mole located on complex surface
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from an outpatient population of subjects at Beckman Laser Medical Clinic, University of California, Irvine.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Changes in human skin structure | up to 12 weeks
  Comparison Imaging Changes in human skin structure Between Spatially Modulated Quantitative Spectroscopy and Skin Spect Dermoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Kelly, MD, Principal Investigator — Beckman Laser Institute, UCI
Locations (1):
- Beckman Laser Institute, Irvine, California, United States